CLINICAL TRIAL: NCT04972630
Title: Implementation of Home-Based Palliative Care in Limited Resource Settings
Brief Title: R21 India Pal-Care Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Tata Medical Center (Other)
Responsible Party: Principal Investigator, Suparna Qanungo, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 00089815; 1R21CA252850-01 (NIH); 2019/GOVT/25/IRB8 (Other: Tata Medical Center, Kolkata, India); 2019-3793 (Other: Indian Council of Medical Research (ICMR), India)
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cancer Palliative Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Control group participants will be recruited from the cancer patients in need of palliative care at Tata Medical Center (TMC), Kolkata, India. Participants will be recruited and consented by TMC researchers. There will be random allocation to the "control" or "Pal-Care" group. The control group (n=45) will receive "usual care" palliative services in which the patient or caregiver (by proxy) must visit the Tata Medical Center (TMC) cancer center for care. TMC services include consultation with a multi-disciplinary team (oncologist, nurse, psychologist), a 21-day morphine supply at reduced cost (as morphine is regulated in use),basic training on medication usage, catheter and wound care, other topics as relevant,and psychological counseling. Patients (or their proxy) must return to the cancer center as needed for follow up care and they are provided a 24/7 hotline to call in case of emergency.
  Interventions: Behavioral: Control-Usual Care
- Pal-Care (Experimental): Intervention group participants will be recruited from cancer patients in need of palliative care at Tata Medical Center (TMC), Kolkata, India. Pal-Care will be delivered over a 6-month period. At baseline visit, the patient and their caregiver will meet with their community health worker (CHW) and clinical team and an individualized care plan will be created. Patients will be assigned to the CHW living nearest to their home. The CHW will make home visits to patients 1+ times weekly, depending on patient need. At each visit, the CHW will use resources from the WHO Palliative Care Toolkit to: 1)monitor patient condition, 2) provide basic palliative care (medication administration, wound care, catheter care), 3) deliver prescribed morphine, 4) teach caregivers to deliver care,5) monitor pain and symptom control, and 6) assist patients to access their oncologists and other resources. Timely communication between CHW and clinical team will be maintained using a tele-health platform.
  Interventions: Behavioral: Pal-Care
- Post-Intervention Interviews (No Intervention): Semi-structured interviews of stakeholder groups will be conducted by MUSC researchers who are well-trained and speak the local language, to evaluate the Pal-Care intervention. We will conduct 20 key informant interviews/KIIs (or until saturation is reached), representing Pal-Care clinical team members, CHWs and patients/caregivers, who participated in the intervention at TMC, India. Clinicians will include social workers, oncology nurses, cancer center administrators, counselors, and palliative care oncologists. Patients/ caregivers will be purposefully selected to represent experiences across different cancers, clinical problems and assigned CHWs. Interviews will be performed in-person or over a telehealth platform, as needed. Interviews will query barriers, facilitators, optimal strategies, experiences, needs and expectations for palliative care delivery. Interviews will be digitally recorded, transcribed and analyzed.

INTERVENTIONS:
Behavioral: Pal-Care — Pal-Care intervention participants will receive a 6-month intervention based upon the WHO toolkit and it will be delivered by the community health workers (CHWs). The goal of this pragmatic clinical trial is to test and evaluate a home-based palliative care intervention for utilizing community health workers to facilitate the delivery of palliative care to cancer patients in rural India. More details provided in the "intervention" arms section. After the intervention, clinicians, CHWs and a purposefully selected set of patients/caregivers, who were involved in the Pal-Care will be interviewed to understand their experiences, needs, expectations, barriers, facilitators and strategies.
  Arms: Pal-Care
Behavioral: Control-Usual Care — The control group will receive "usual care" palliative services in which the patient or caregiver (by proxy) must visit the Tata Medical Center (TMC) cancer center for care. TMC services include consultation with a multi-disciplinary team (oncologist, nurse, psychologist), a 21-day morphine supply at reduced cost (as morphine is regulated in use),basic training on medication usage, catheter and wound care, other topics as relevant,and psychological counseling. Patients (or their proxy) must return to the cancer center as needed for follow up care and they are provided a 24/7 hotline to call in case of emergency.
  Arms: Control

SUMMARY:
The goal of this pragmatic clinical trial is to test and evaluate a home-based palliative care intervention for utilizing community health workers to facilitate the delivery of palliative care to cancer patients in rural India. The study builds upon use of the World Health Organization-endorsed "Palliative Care Toolkit," which provides a comprehensive suite of evidence-based materials for delivering palliative care in limited resource settings. For the intervention, two specific aims will be addressed to evaluate: 1) implementation of the intervention within the context of the RE-AIM Framework and 2) outcomes of this intervention to determine its relative effects compared to a standard control group on patients' palliative care needs, symptom burden, quality of life (QOL) and experience with care.

DETAILED DESCRIPTION:
This pragmatic clinical trial is a collaboration between the Medical University of South Carolina (MUSC)and Tata Medical Center (TMC), a cancer center in Kolkata, India. The study has two parts: a) Implementation of a Pal-Care intervention as compared to control/no intervention b) Qualitative post-intervention evaluation.

The part a) of the study is conducted at Tata Medical Center (TMC) in Kolkata, India, under the supervision of the site PI, Dr. Gaurav Kumar. All participants will be recruited from among the TMC patients who are referred to cancer palliative care and will be grouped to the "Control" or "Pal-Care" intervention groups. This part of the study will compare an intervention group of patients who will receive home-based palliative services (Pal-Care)from community health workers (CHWs) vs. a control group of patients who will receive cancer-center based palliative services. This intervention implementation part of the study is approved by TMC Ethics Board and Indian Council of Medical Research (ICMR), approval letter on file with MUSC IRB. MUSC relies on TMC IRB for this part and the ICF document is approved by the TMC Ethics Board in India.

The part b) of the study (under purview of MUSC IRB) involves post-intervention qualitative interviews. MUSC research team will evaluate the implementation and effect of the Pal-Care intervention to deliver CHW navigated home-based palliative care for rural cancer patients in India. The participants of this part of the study will also be from India and include stakeholders, representing all Pal-Care clinical team members and CHWs and patients/caregivers who participated in the Pal-Care intervention. This part has a waiver of signed consent.

The RE-AIM framework guides our evaluation plan to measure the reach, effectiveness, adoption, implementation and maintenance of the Pal-Care intervention. Diverse data sources will be used to evaluate the intervention within the REAIM Framework.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 years and over, any cancer type, late state cancer, residence in 24 Parganas Region, West Bengal, India, physician documentation in medical record that patient is to receive palliative care, patient willingness to participate in data collection.

Exclusion Criteria:

* Prisoner; diagnoses of substance addiction (illicit drugs), Mentally unstable or having moderate to severe mental health issue or incapable of decision making, Unable to speak or communicate with ease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suparna Qanungo, PhD, Principal Investigator — Associate Professor
Locations (1):
- Tata Medical Center, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: No
MUSC researchers have access to ONLY de-identified data. All source documents and identifiers are with Dr. Gaurav Kumar, Site PI at TATA Medical Centre, Rajarhat, Kolkata, India

REFERENCES:
- [Derived] Qanungo S, Cartmell KB, Mueller M, Butcher M, Sarkar S, Carlson TG, Madisetti M, Kumar G. Comparison of home-based palliative care delivered by community health workers versus usual care: research protocol for a pilot randomized controlled trial. BMC Palliat Care. 2023 Sep 2;22(1):125. doi: 10.1186/s12904-023-01235-z. PMID 37658397
- See also: Comparison of home-based palliative care delivered by community health workers versus usual care: research protocol for a pilot randomized controlled trial (PMID 37658397) — https://pubmed.ncbi.nlm.nih.gov/37658397/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Post-intervention interviews: The participants were people who had in some way engaged in the Pal-Care intervention as a provider, community health worker or patient. Hence for the research purpose, we only needed to know if they had engaged in the intervention and NO additional demographics/OUTCOME DATA were counted twice for research.
  All participants were informed through a statement of research (waiver of signed consent in place) and verbally consented prior to conducting interviews.
Groups:
- Post-Intervention Interviews: Semi-structured interviews of stakeholder groups will be conducted by MUSC researchers who are well-trained and speak the local language, to evaluate the Pal-Care intervention. We will conduct 20 key informant interviews/KIIs (or until saturation is reached), representing Pal-Care clinical team members, CHWs and patients/caregivers, who participated in the intervention at TMC, India. The patients were a part of the intervention group. Clinicians will include social workers, oncology nurses, cancer center administrators, counselors, and palliative care oncologists. Patients/ caregivers will be purposefully selected to represent experiences across different cancers, clinical problems and assigned CHWs. Interviews will be performed in-person or over a telehealth platform, as needed. Interviews will query barriers, facilitators, optimal strategies, experiences, needs and expectations for palliative care delivery. Interviews will be digitally recorded, transcribed and analyzed.
Period: Overall Study
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Started | 45 | 45 | 22
Completed | 8 | 8 | 22
Not Completed | 37 | 37 | 0
Not completed — Death due to disease progression, lost to follow-up, consent withdrawal | 37 | 37 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was only meant to be collected for control and intervention participants. For the post-intervention interviews, the participants were people who had in some way engaged in the Pal-Care intervention as a provider, community health worker or patient. Hence for the research purpose, we are not double counting as the outcome data is only reflective of control and intervention groups and not impacted by the qualitative interviews.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Pal-Care | Post-Intervention Interviews | Total
Number analyzed (Participants) | 43 | 43 | 22 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  years
    number analyzed (Participants) | 43 | 43 | 00 | 86
    (all) | 59.8 (12.8) | 60.4 (15.9) |  | 60.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    number analyzed (Participants) | 43 | 43 | 0 | 86
    Female | 20 | 19 | 0 | 39
    Male | 23 | 24 | 0 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    number analyzed (Participants) | 43 | 43 | 0 | 86
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 43 | 43 | 0 | 86
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    India: number analyzed (Participants) | 43 | 43 | 0 | 86
    India | 43 | 43 | 0 | 86
Marital Status [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Single: number analyzed (Participants) | 43 | 43 | 00 | 86
    Single | 0 | 2 |  | 2
    Married: number analyzed (Participants) | 43 | 43 | 00 | 86
    Married | 36 | 29 |  | 65
    Widowed: number analyzed (Participants) | 43 | 43 | 00 | 86
    Widowed | 7 | 12 |  | 19
Religion [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Hindu: number analyzed (Participants) | 43 | 43 | 00 | 86
    Hindu | 36 | 35 |  | 71
    Muslim: number analyzed (Participants) | 43 | 43 | 00 | 86
    Muslim | 5 | 8 |  | 13
    Christian: number analyzed (Participants) | 43 | 43 | 00 | 86
    Christian | 2 | 0 |  | 2
Highest level of education completed [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Less than high school degree: number analyzed (Participants) | 43 | 43 | 00 | 86
    Less than high school degree | 5 | 7 |  | 12
    High school degree: number analyzed (Participants) | 43 | 43 | 00 | 86
    High school degree | 16 | 18 |  | 34
    Some college but no degree: number analyzed (Participants) | 43 | 43 | 00 | 86
    Some college but no degree | 1 | 0 |  | 1
    Bachelor degree (B.S, B.A, B.Com etc.): number analyzed (Participants) | 43 | 43 | 00 | 86
    Bachelor degree (B.S, B.A, B.Com etc.) | 17 | 16 |  | 33
    Master's degree or above: number analyzed (Participants) | 43 | 43 | 00 | 86
    Master's degree or above | 4 | 1 |  | 5
    Prefer not to answer: number analyzed (Participants) | 43 | 43 | 00 | 86
    Prefer not to answer | 0 | 1 |  | 1
Employment status [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Employed with an organization: number analyzed (Participants) | 43 | 43 | 00 | 86
    Employed with an organization | 0 | 1 |  | 1
    Self-Employed: number analyzed (Participants) | 43 | 43 | 00 | 86
    Self-Employed | 4 | 4 |  | 8
    Not employed, looking for work: number analyzed (Participants) | 43 | 43 | 00 | 86
    Not employed, looking for work | 1 | 0 |  | 1
    Not employed, NOT looking for work: number analyzed (Participants) | 43 | 43 | 00 | 86
    Not employed, NOT looking for work | 16 | 13 |  | 29
    Retired: number analyzed (Participants) | 43 | 43 | 00 | 86
    Retired | 10 | 13 |  | 23
    Disabled, not able to work: number analyzed (Participants) | 43 | 43 | 00 | 86
    Disabled, not able to work | 12 | 11 |  | 23
    Prefer not to answer: number analyzed (Participants) | 43 | 43 | 00 | 86
    Prefer not to answer | 0 | 1 |  | 1
Income [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Less than INR 5,000: number analyzed (Participants) | 43 | 43 | 00 | 86
    Less than INR 5,000 | 0 | 3 |  | 3
    INR 5,000 to INR 24,999: number analyzed (Participants) | 43 | 43 | 00 | 86
    INR 5,000 to INR 24,999 | 17 | 17 |  | 34
    INR 25,000 to INR 49,999: number analyzed (Participants) | 43 | 43 | 00 | 86
    INR 25,000 to INR 49,999 | 12 | 9 |  | 21
    INR 50,000 to INR 99,999: number analyzed (Participants) | 43 | 43 | 00 | 86
    INR 50,000 to INR 99,999 | 7 | 4 |  | 11
    INR100, 000 (1 lacs) or more: number analyzed (Participants) | 43 | 43 | 00 | 86
    INR100, 000 (1 lacs) or more | 2 | 7 |  | 9
    Prefer not to answer: number analyzed (Participants) | 43 | 43 | 00 | 86
    Prefer not to answer | 5 | 3 |  | 8
Living location [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Rural village: number analyzed (Participants) | 43 | 43 | 00 | 86
    Rural village | 10 | 12 |  | 22
    Suburban town: number analyzed (Participants) | 43 | 43 | 00 | 86
    Suburban town | 11 | 10 |  | 21
    Urban city: number analyzed (Participants) | 43 | 43 | 00 | 86
    Urban city | 22 | 21 |  | 43
Members in household (including self) [Mean (Standard Deviation); unit: Members in household (including self)] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Members in household (including self)
    number analyzed (Participants) | 43 | 43 | 00 | 86
    (all) | 4.8 (2.4) | 4.5 (2.8) |  | 4.7 (2.6)
Number of dependents in family [Mean (Standard Deviation); unit: Number of dependents in family] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Number of dependents in family
    number analyzed (Participants) | 43 | 43 | 00 | 86
    (all) | 2.8 (1.6) | 2.7 (2.3) |  | 2.7 (1.95)
Relationship with primary caregiver [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Parent: number analyzed (Participants) | 43 | 43 | 00 | 86
    Parent | 0 | 2 |  | 2
    Spouse: number analyzed (Participants) | 43 | 43 | 00 | 86
    Spouse | 25 | 18 |  | 43
    Sibling: number analyzed (Participants) | 43 | 43 | 00 | 86
    Sibling | 0 | 1 |  | 1
    Other: number analyzed (Participants) | 43 | 43 | 00 | 86
    Other | 18 | 22 |  | 40
Has health insurance or funds [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    number analyzed (Participants) | 43 | 43 | 00 | 86
    Yes | 20 | 15 |  | 35
    No | 23 | 28 |  | 51
Health insurance [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Governmental insurance: number analyzed (Participants) | 43 | 43 | 00 | 86
    Governmental insurance | 4 | 5 |  | 9
    Private insurance: number analyzed (Participants) | 43 | 43 | 00 | 86
    Private insurance | 16 | 10 |  | 26
    Self-pay: number analyzed (Participants) | 43 | 43 | 00 | 86
    Self-pay | 23 | 28 |  | 51
Diagnosis based on system [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Breast: number analyzed (Participants) | 43 | 43 | 00 | 86
    Breast | 4 | 5 |  | 9
    Cancer of Unknown Primary (CUP): number analyzed (Participants) | 43 | 43 | 00 | 86
    Cancer of Unknown Primary (CUP) | 1 | 1 |  | 2
    Genitourinary: number analyzed (Participants) | 43 | 43 | 00 | 86
    Genitourinary | 2 | 2 |  | 4
    GI Cancers: number analyzed (Participants) | 43 | 43 | 00 | 86
    GI Cancers | 19 | 13 |  | 32
    Gynecological: number analyzed (Participants) | 43 | 43 | 00 | 86
    Gynecological | 6 | 8 |  | 14
    Head & Neck: number analyzed (Participants) | 43 | 43 | 00 | 86
    Head & Neck | 6 | 4 |  | 10
    Skin: number analyzed (Participants) | 43 | 43 | 00 | 86
    Skin | 1 | 0 |  | 1
    Thoracic: number analyzed (Participants) | 43 | 43 | 00 | 86
    Thoracic | 4 | 10 |  | 14
Body weight (kg) [Mean (Standard Deviation); unit: kg] — Population: One patient in the "control" group could not be mobilized at the point of time, hence weight could not be taken.
  Additionally, baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  kg
    number analyzed (Participants) | 41 | 42 | 00 | 83
    (all) | 57.8 (13.6) | 57.8 (12.9) |  | 57.8 (13.2)
Has reliable internet access [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    number analyzed (Participants) | 43 | 43 | 00 | 86
    Yes | 43 | 40 |  | 83
    No | 0 | 3 |  | 3
Comfortable using [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Computers: number analyzed (Participants) | 43 | 43 | 00 | 86
    Computers | 7 | 2 |  | 9
    iPad/tablet: number analyzed (Participants) | 43 | 43 | 00 | 86
    iPad/tablet | 2 | 2 |  | 4
    Smartphone: number analyzed (Participants) | 43 | 43 | 00 | 86
    Smartphone | 33 | 36 |  | 69
    None: number analyzed (Participants) | 43 | 43 | 00 | 86
    None | 1 | 3 |  | 4
ECOG status [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Well: number analyzed (Participants) | 43 | 43 | 00 | 86
    Well | 2 | 2 |  | 4
    Active - able to do light work: number analyzed (Participants) | 43 | 43 | 00 | 86
    Active - able to do light work | 11 | 14 |  | 25
    Self-caring - but unable to work: number analyzed (Participants) | 43 | 43 | 00 | 86
    Self-caring - but unable to work | 19 | 22 |  | 41
    Bedridden >50% of the day: number analyzed (Participants) | 43 | 43 | 00 | 86
    Bedridden >50% of the day | 11 | 5 |  | 16
Problems at identified at enrollment [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    Emotional issues: number analyzed (Participants) | 43 | 43 | 00 | 86
    Emotional issues | 30 | 34 |  | 64
    Spiritual issues: number analyzed (Participants) | 43 | 43 | 00 | 86
    Spiritual issues | 18 | 16 |  | 34
    Social issues: number analyzed (Participants) | 43 | 43 | 00 | 86
    Social issues | 32 | 30 |  | 62
Discussion of non-escalation [Count of Participants; unit: Participants] — Population: Baseline data was only meant to be collected for control and intervention participants. Hence no baseline information was collected for interview participants.
  Participants
    number analyzed (Participants) | 43 | 43 | 00 | 86
    Yes | 21 | 18 |  | 39
    No | 22 | 25 |  | 47

OUTCOME MEASURES:

1. Primary Outcome: Palliative Care Outcomes (POS Total Scores)
Description: Multidimensional palliative care outcomes will be measured with Palliative Care Outcomes (POS) Scale that measures physical and psychological symptoms; spiritual, practical and emotional concerns; and psychosocial needs of patient/family. The overall POS scale included 10 items, it is a 5-point Likert scale, scored from 0 to 4, with a total summed score ranging from 0-40. A score of 0 indicates that the particular issue is not a problem at all and a score of 4 indicates that the issue is an overwhelming burden/concern for the patient. The higher the total score, the worser the palliative care outcomes are.
Time Frame: 6-month
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 43 | 43 | 0
score on a scale
  Baseline | 23.5 [18.7 to 28.3] | 22.9 [18.1 to 27.7] |
  Week 4: number analyzed (Participants) | 31 | 29 | 0
  Week 4 | 22.2 [16.9 to 27.5] | 22.1 [15.9 to 28.3] |
  Week 12: number analyzed (Participants) | 20 | 13 | 0
  Week 12 | 22.1 [16.9 to 27.3] | 20.8 [15 to 26.6] |
  Week 24: number analyzed (Participants) | 8 | 8 | 0
  Week 24 | 21.3 [15.1 to 27.5] | 19.4 [12.4 to 26.4] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Baseline control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 0.6
Statistical Analysis 2: Comparison: Control vs Pal-Care; Week 4 control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 0.1
Statistical Analysis 3: Comparison: Control vs Pal-Care; Week 12, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 1.3
Statistical Analysis 4: Comparison: Control vs Pal-Care; Week 24, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 1.9

2. Primary Outcome: Average Score for Quality of Life (QOL) Physical Domain
Description: Quality of Life will be will be assessed with the 26-item WHOQOL-BREF(WHO-Quality of life-BREFF) Scale that addresses 4 QOL domains (physical, psychological, social relationships and environment. The Quality of Life (QOL) Physical Domain scale included 7 items, it is a 5-point Likert scale, scored from 0 to 4, summed over the 7 domain items multiplied by 4, transformed to a 0-100 scale using the formula (score-4)x(100/16). A score of 0 indicates the poorest level for physical QOL and a score of 4 indicates that the highest level of physical QOL for the patient. Higher total score indicates better physical QOL for the patient.
Time Frame: Baseline to Week 4
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 31 | 29 | 0
score on a scale | 55.6 [35.7 to 75.5] | 56.1 [43.1 to 69.1] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 0.5

3. Primary Outcome: Average Score for Quality of Life (QOL) Physical Domain
Description: as for outcome 2
Time Frame: Week 4
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 31 | 29 | 0
score on a scale | 51.3 [30.4 to 72.2] | 52.8 [32.1 to 73.5] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 1.5

4. Primary Outcome: Average Score for Quality of Life (QOL) Physical Domain
Description: as for outcome 2
Time Frame: Baseline to Week 12
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 20 | 13 | 0
score on a scale | 59.1 [42 to 76.2] | 57.4 [44.3 to 70.5] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -1.7

5. Primary Outcome: Average Score for Quality of Life (QOL) Physical Domain
Description: as for outcome 2
Time Frame: Week 12
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 20 | 13 | 0
score on a scale | 55.6 [33.1 to 78.1] | 52.8 [34.5 to 71.1] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -2.8

6. Primary Outcome: Average Score for Quality of Life (QOL) Physical Domain
Description: as for outcome 2
Time Frame: Baseline to Week 24
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 8 | 8 | 0
score on a scale | 69.4 [58.4 to 80.4] | 60.2 [52.1 to 68.3] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -9.2

7. Primary Outcome: Average Score for Quality of Life (QOL) Physical Domain
Description: as for outcome 2
Time Frame: Week 24
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 8 | 8 | 0
score on a scale | 59.7 [33.4 to 86] | 62.9 [40.1 to 85.7] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 3.2

8. Primary Outcome: Average Score for Quality of Life (QOL) Psychological Domain
Description: Quality of Life will be will be assessed with the 26-item WHOQOL-BREF(WHO-Quality of life-BREFF) Scale that addresses 4 QOL domains (physical, psychological, social relationships and environment. The Quality of Life (QOL) Psychological Domain scale included 6 items, it is a 5-point Likert scale, scored from 0 to 4, summed over the 6 domain items multiplied by 4, transformed to a 0-100 scale using the formula (score-4)x(100/16). A score of 0 indicates the poorest level for psychological QOL and a score of 4 indicates that the highest level of psychological QOL for the patient. Higher total score indicates better psychological QOL for the patient.
Time Frame: Baseline to Week 4
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 31 | 29 | 0
score on a scale | 63.3 [44.8 to 81.8] | 58.3 [42.2 to 74.4] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -5

9. Primary Outcome: Average Score for Quality of Life (QOL) Psychological Domain
Description: as for outcome 8
Time Frame: Week 4
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 31 | 29 | 0
score on a scale | 58.2 [42.2 to 74.2] | 53.7 [30.3 to 77.1] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -4.5

10. Primary Outcome: Average Score for Quality of Life (QOL) Psychological Domain
Description: as for outcome 8
Time Frame: Baseline to Week 12
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 20 | 13 | 0
score on a scale | 67.3 [50.4 to 84.2] | 60.9 [45 to 76.8] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -6.4

11. Primary Outcome: Average Score for Quality of Life (QOL) Psychological Domain
Description: as for outcome 8
Time Frame: Week 12
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 20 | 13 | 0
score on a scale | 59.6 [38.6 to 80.6] | 55.8 [39.6 to 72] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -3.8

12. Primary Outcome: Average Score for Quality of Life (QOL) Psychological Domain
Description: as for outcome 8
Time Frame: Baseline to Week 24
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 8 | 8 | 0
score on a scale | 76.6 [60 to 93.2] | 59.9 [47.7 to 72.1] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -16.7

13. Primary Outcome: Average Score for Quality of Life (QOL) Psychological Domain
Description: as for outcome 8
Time Frame: Week 24
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 8 | 8 | 0
score on a scale | 62.0 [39.4 to 84.6] | 62.5 [39.2 to 85.8] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 0.5

14. Primary Outcome: Total Score for Quality of Life (QOL) Social Domain
Description: Quality of Life will be will be assessed with the 26-item WHOQOL-BREF(WHO-Quality of life-BREFF) Scale that addresses 4 QOL domains (physical, psychological, social relationships and environment. The Quality of Life (QOL) Social Domain scale included 3 items, it is a 5-point Likert scale, scored from 0 to 4, summed over the 3 domain items multiplied by 4, transformed to a 0-100 scale using the formula (score-4)x(100/16). A score of 0 indicates the poorest level for social QOL and a score of 4 indicates that the highest level of social QOL for the patient. Higher total score indicates better social QOL for the patient.
Time Frame: 6 months
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 43 | 43 | 0
score on a scale
  Baseline | 81.1 [61.7 to 100.5] | 81.5 [64.4 to 98.6] |
  Week 4: number analyzed (Participants) | 31 | 29 | 0
  Week 4 | 73.3 [50.1 to 96.5] | 78.7 [59.8 to 97.6] |
  Week 12: number analyzed (Participants) | 20 | 13 | 0
  Week 12 | 77.9 [52.4 to 103.4] | 78.8 [61.6 to 96] |
  Week 24: number analyzed (Participants) | 8 | 8 | 0
  Week 24 | 80.2 [58.5 to 101.9] | 82.8 [65.2 to 100.4] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Baseline, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 0.4
Statistical Analysis 2: Comparison: Control vs Pal-Care; Week 4, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 5.5
Statistical Analysis 3: Comparison: Control vs Pal-Care; Week 12, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 0.9
Statistical Analysis 4: Comparison: Control vs Pal-Care; Week 24, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 2.6

15. Primary Outcome: Total Score for Quality of Life (QOL) Environment Domain
Description: Quality of Life will be will be assessed with the 26-item WHOQOL-BREF(WHO-Quality of life-BREFF) Scale that addresses 4 QOL domains (physical, psychological, social relationships and environment. The Quality of Life (QOL) Environmental Domain scale included 8 items, it is a 5-point Likert scale, scored from 0 to 4, summed over the 8 domain items multiplied by 4, transformed to a 0-100 scale using the formula (score-4)x(100/16). A score of 0 indicates the poorest level for environmental QOL and a score of 4 indicates that the highest level of environmental QOL for the patient. Higher total score indicates better environmental QOL for the patient.
Time Frame: 6 Months
Population: Outcome surveys/data collection were not conducted on Post-intervention interview participants
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
Number analyzed (Participants) | 43 | 43 | 0
score on a scale
  Baseline | 68.6 [55.1 to 82.1] | 66.4 [53.1 to 79.7] |
  Week 4: number analyzed (Participants) | 31 | 29 | 0
  Week 4 | 65.8 [53.5 to 78.1] | 66.4 [49.7 to 83.1] |
  Week 12: number analyzed (Participants) | 20 | 13 | 0
  Week 12 | 67.1 [53.3 to 80.9] | 66.1 [51.7 to 80.5] |
  Week 24: number analyzed (Participants) | 8 | 8 | 0
  Week 24 | 72.7 [59.5 to 85.9] | 71.9 [52.2 to 91.6] |
Statistical Analysis 1: Comparison: Control vs Pal-Care; Baseline, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -2.2
Statistical Analysis 2: Comparison: Control vs Pal-Care; Week 4, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = 0.5
Statistical Analysis 3: Comparison: Control vs Pal-Care; Week 12, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -0.9
Statistical Analysis 4: Comparison: Control vs Pal-Care; Week 24, control vs. intervention; Test type: Other — Comparison via 95% confidence interval; Mean Difference (Final Values) = -0.8

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks
Description: SAEs (patients could have more than 1 SAE, therefor does not add to total N of patients)
  All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed for the "Post-Intervention Interviews" Arm/Group.
Arm/Group | Control | Pal-Care | Post-Intervention Interviews
All-Cause Mortality (participants affected / at risk) | 17/43 | 18/43 | 0/0
Serious Adverse Events (participants affected / at risk) | 19/43 | 24/43 | 0/0
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=43) | Pal-Care (N=43) | Post-Intervention Interviews (N=0)
Consumption of a liquid mosquito repellent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — Consumption of a liquid mosquito repellent. Volume not specified. C/o mild SOB. No other complain.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Shortness of breath.
Progression of Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Breathlessness, cold, reduced intake of food.
Progression of Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Breathlessness, Urinary retention.
Progression of Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Respiratory distress.
Progression of Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Shortness of breath, chest pain, disorientation.
Progression of Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Constipation, nausea, abdominal distension and pain, vomiting.
Progression of Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Shortness of breath
Progression of Disease (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — Anorexia, not able to eat or drink, high colored urine, yellowish discoloration, generalized itching.
Progression of Disease (General disorders) | 0 (0) | 1 (1) | 0 (0) — Both leg pedal edema, abdominal distension, generalized weakness.
Progression of Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Shortness of breath.
Dyselectrolytemia and Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Drowsiness and disorientation with vomiting.
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Epigastric pain, petechial lesion in the right forearm.
Progression of Disease (General disorders) | 1 (1) | 0 (0) | 0 (0) — Abdominal distention, Shortness of breath, seizures, senselessness, fever and coffee colored stool.
Subacute intestinal obstruction. (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Abdominal pain, abdominal tightness, bloating, dyspepsia, anorexia, generalized weakness, vomiting (brownish color).
Subacute intestinal obstruction. (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Abdominal pain.
Progression of disease and Dyselectrolytemia (General disorders) | 1 (1) | 0 (0) | 0 (0) — Abdominal discomfort and pain, decreased urine output and irrelevant talks
Infection and Dyselectrolytemia (General disorders) | 0 (0) | 1 (1) | 0 (0) — Abdominal distension, Weakness ,Vomiting.
Disorientation and Reduced intake of Food (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) — Bleeding from lower lip, disorientation on and off, reduced intake of food, generalized weakness.
Progression of Disease (General disorders) | 1 (1) | 0 (0) | 0 (0) — Breathlessness on exertion, Anasarca
Ulcer proliferative Lesion (General disorders) | 0 (0) | 1 (1) | 0 (0) — Bleeding and headache. On examination he was found to have a large ulcer proliferative lesion in his left cheek and angle of mouth. The lesion was bleeding and pus was draining which was foul-smelling.
Hypertension, Dehydrated, Cachectic, and Tense Ascites (General disorders) | 0 (0) | 1 (1) | 0 (0) — Drowsiness, generalized weakness and abdominal distension. Hypotension with a BP of 70/40mmHg and dehydrated and cachectic and also had tense ascites.
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Dysphagia, anorexia, generalized weakness.
Sepsis and Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Generalized weakness, loose stool, constipation, generalized body pain, appetite loss.
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Generalized weakness, Insomnia and Anxiety.
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Generalized weakness, Black stools
Fluctuating BP and blood sugar (General disorders) | 0 (0) | 1 (1) | 0 (0) — Generalized weakness, fluctuating BP and blood sugar, occasional bleeding from tumor site, dehydration.
Sepsis, Diabetic Ketoacidosis and Dyselectrolytemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Generalized weakness, decreased intake of food
Low hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Bleeding per rectum and vagina.
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Breathlessness intermittently, Bleeding PV, Recto-vaginal fistula, Feverish.
Hypercalcemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Constipation, anorexia and weakness.
Dyselectrolytemia and Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Drowsiness and constipation, decreased intake of food.
Progression of Disease and Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Drowsiness, No urine.
Progression of Disease (General disorders) | 2 (2) | 0 (0) | 0 (0) — Unresponsive.
Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Vomiting, generalized weakness and abdominal pain.
Chest Infection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Shortness of breath, hypotension.
Deep Vein Thrombosis, Dyselectrolytemia, and Suspected Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Swelling of right upper limbs, generalized weakness and tremors ,deep vein thrombosis, Dyselectrolytemia and suspected sepsis
Progression Of Disease With Pneumonia (General disorders) | 1 (1) | 0 (0) | 0 (0) — Vomiting, Dizziness, Blurring of vision, Headache, Cough and Back pain.
Dyselectrolytemia and Sepsis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Shortness of breath, generalized weakness.
Hypoproteinemia, Anemia and Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Dysuria, scrotal swelling in genital area and whole body edema, hypotensive
Chickenpox (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Fever with rash.
Cerebral metastases (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Involuntary facial muscle twitching, restlessness, drowsiness, back pain, seizures.
Electrolyte disturbance. (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — Mild facial deviation. Face deviated toward one side for 5 sec, and there was dribbling of water from angle of mouth.
Dyselectrolytemia and Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Reduced appetite, unable to swallow, Imbalance in gait, Urinary incontinence, Drowsy, Loose stools.
ICD Block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — No output from ICD.
Sepsis and Hypoglycemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Respiratory distress, slurring of speech.
Sepsis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Drowsiness.
Infection and UTI (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Fever and weakness.
Upper GI bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Hematemesis
Progression of Disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Pain in abdomen & vomiting.
Hypogastric plexus and Block (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Pain in lower abdomen and left leg.
Cancer Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — Pain, cough, low grade fever.
PR Bleeding and Generalized weakness (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — PR Bleeding, Leading to anemia, Malena, Generalized weakness.
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Severe respiratory distress, tachycardia, hyperglycemia.
severe anemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Shortness of breath
Progression of Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Shortness of breath, Hemoptysis, Melena, Upper abdomen pain, Vomiting, jaundice
Progression of Disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Tumor site bleeding, Shortness of breath.
Patient Expired at Home (General disorders) | 16 (16) | 14 (14) | 0 (0) — Family informed that patient expired at home.
Patient Expired at Local Hospital (General disorders) | 1 (1) | 4 (4) | 0 (0) — Family informed that patient expired at local Hospital.
Progression of Disease (General disorders) | 1 (1) | 0 (0) | 0 (0) — Patient came in emergency with c/o twitching of right side face, pain in right side chest, edema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT04972630/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT04972630/SAP_001.pdf
  • Informed Consent Form (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT04972630/ICF_002.pdf